CLINICAL TRIAL: NCT06910696
Title: Erector Spinae Plane Block Versus Modified Thoracolumbar Interfascial Plane Block for Rapid Recovery and Rehabilitation After Lumber Discectomy: A Randomized Study
Brief Title: Erector Spinae Plane Block Versus Modified Thoracolumbar Interfascial Plane Block
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Mohamed Medhat, assistant professor of anesthesia and surgical intensive care (Principal Investigator), Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZU-IRB#1074/25-Feb-2025
Record Dates: First submitted 2025-03-19; First posted 2025-04-04 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Achievement of High-quality Analgesia, Rapid Recovery With Rehabilitation in Lumber Spine Discectomy
Keywords: erector spinae plane block modified thoracolumbar interfascial plane block perioperative analgesia lumber spine discectomy?

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- • Control Group (No Intervention): Patients will receive standard analgesia (paracetamol 15mg/kg plus fentanyl 1ug/kg) iv.
- (mTLIP )Group (Active Comparator): Patients will receive 20 mL of 0.25% bupivacaine on each side through Modified thoracolumbar interfascial block
  Interventions: Drug: Regional Anesthetic Injection
- (ESPB) Group (Active Comparator): Patients will receive 20 mL of 0.25% bupivacaine on each side through Erector spinae block
  Interventions: Drug: Regional Anesthetic Injection

INTERVENTIONS:
Drug: Regional Anesthetic Injection — The probe will be placed in the parasagittal plane at the level of the L3 vertebrae. The spinous process will be visualized, and the probe was moved 3 cm laterally from the midline. The erector spinae musclewill be visualized above the transverse process. The needle will be punctured in the craniocaudal direction using the in-plane technique. The needle will be directed superior to the transverse process . Then, 2 mL normal saline solution will be injected into the deep fascia of the erector spinae muscle to confirm the proper injection site. After ensuring the location of the needle, 20 mL of 0.25% bupivacaine will be administered. The same ESPB procedure will be performed on the other side. In total, 40 mL of 0.25% bupivacaine was administered
  Arms: (ESPB) Group
Drug: Regional Anesthetic Injection — The probe will be placed vertically at the L3 vertebrae level. The spinous process and the interspinous muscles (i.e., multifidus, longissimus, and iliocostalis) will be visualized as the anatomic guide points. The probewill be moved laterally to identify the longissimus and iliocostalis muscles . The needlewill be inserted between the longissimus and iliocostalis in the medial-to-lateral direction using the in-plane technique. After confirming the location of the needle, 20 mL of 0.25% bupivacaine will be administered. The same mTLIP procedure will be performed on the opposite side. In total, 40 mL of 0.25% bupivacaine will be administered
  Arms: (mTLIP )Group

SUMMARY:
the purpose of this study is to compare of better postoperative analgesia following lumber spine discectomy

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient.
* Physical status: ASA 1& II.
* BMI = (25-30 kg/m2).
* Type of operation: elective Lumbar discectomy .

Exclusion Criteria:

* Altered mental state.
* Patients with known history of allergy to study drugs.
* Advanced hepatic, renal, cardiovascular, and respiratory diseases.
* Patients with chronic pain.
* Patients receiving anticoagulants.
* Contraindications of regional anesthesia, e.g., allergy to local anesthetics, coagulopathy, or septic focus at site of injection.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | up to 1 weak postoperative.
  from the day of admission till discharge from hospital

SECONDARY OUTCOMES:
The recovery time | up to 30 minutes postoperative.
  time from discontinuation of isoflurane to first response to verbal command
The time of discharge | up to 2 hours postoperative.
  The time from arrival to the PACU to discharge to the ward
6 minutes walk test | 24 hours postoperative
  involves walking for 6 min on a 30 m walking path and measuring the distance
Functional reach test | 24 hours postoperative
  quantifies participants' dynamic in-place standing balance control to reach distance. The distance between the starting and maximal forward reach distance beyond the participant's arm length represents the reach distance and is recorded in centimeters
Time up and go test | 24 hours postoperative
  objective measure of functional disability that can be used to evaluate various activities such as standing, accelerating, walking, decelerating, and turning, which are often limited in patients with lumbar degenerative diseases
Pain intensity | 30 minutes after the end of the surgery, as well as 3, 6, 12, and 24 hours postoperatively
  10-point NRS [(0 = no pain, 10 = worst imaginable pain), 1 - 3: Mild pain (nagging, annoying, slightly interfering with activities of daily living (ADLs), 4 - 6: Moderate pain (significantly interfering with ADLs, 7 - 10: Severe pain (disabling, unable to perform ADLs)]
Time to first call analgesia | 24 hours postoperative
Total naluphine consumption | 24 hours post-operative

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine,zagazig university Egypt Ext. 002 K.Howida@yahoo.com, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: https://pubmed.ncbi.nlm.nih.gov/29318534/ — https://pubmed.ncbi.nlm.nih.gov/29318534/